CLINICAL TRIAL: NCT04386694
Title: Is Photobiomodulation Therapy (PBMT) Combined With Static Magnetic Field (sMF) Able to Decrease the Intensive Care Unit (ICU) Length of Stay for Patients With COVID-19?
Brief Title: Photobiomodulation Therapy Combined With Static Magnetic Field in Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Hospital Tacchini/RS (Unknown)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Full professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3.985.226
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: COVID-19; Respiratory Failure
Keywords: Photobiomodulation Therapy; Static Magnetic Fields; Low-Level Laser Therapy; COVID-19; Invasive Mechanical Ventilation; Respiratory Muscles; Intensive Care United
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A researcher will program the device (PMBT/sMF or placebo) and will be instructed not to inform the patients or other researchers as to the type of treatment (PMBT/sMF or placebo). Therefore, the therapist responsible for the treatment, the investigators and the outcome assessors will be blinded to the type of treatment being administered to the patients. The sounds and signals emitted from the device as well as the information displayed on the screen will be identical, regardless of the type of treatment (PBMT/sMF or placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PBMT/sMF (Experimental): Active PBMT/sMF will be applied once a day, during the ICU stay, until discharge or death. The patients will receive standard physical therapy care associated with PBMT/sMF.
  PBMT/sMF will be applied using MR5™ ACTIV PRO LaserShower, manufactured by Multi Radiance Medical (Solon, OH, USA). This device has 4 diodes of 905 nm (1.25 mW each diode, 0.32 cm2 each), 8 diodes of 633 nm (25 mW each diode, 0.85 cm2 - each), and 8 diodes of 850 nm (40 mW each diode, 0.56 cm2 - each). The static magnetic field is 110 mT.
  Interventions: Device: Active PBMT/sMF
- Placebo PBMT/sMF (Placebo Comparator): Placebo PBMT/sMF will be applied once a day, during the ICU stay, until discharge or death. The patients will receive standard physical therapy care associated with placebo PBMT/sMF.
  The placebo PBMT will be applied using MR5™ ACTIV PRO LaserShower Laser Therapy System, manufactured by Multi Radiance Medical (Solon, OH, USA). The ACTIV PRO emits 905nm, and 850nm via an electric diode energy source with outputs to 0%. The static magnetic field will be also turned off. The 660nm light via an electric diode energy source with outputs to >1% to appear like the active comparator.
  Interventions: Device: Placebo PBMT/sMF

INTERVENTIONS:
Device: Active PBMT/sMF — The PBMT/sMF will be irradiated in the lower thorax and neck areas, with the patients in supine position. PBMT/sMF application time will be 60 seconds per site. The dose used in the lower thorax will be 31.50 J per site, a total of 6 sites will be irradiated, totalizing a dose of 189J. In addition, the dose used in the neck area (bilaterally) will be 31.50J per site, a total of 1 site (bilaterally) will be irradiated, totalizing a dose of 31.50J (bilaterally). PBMT/sMF will be applied using the direct contact method with light pressure on the skin.
  Arms: PBMT/sMF
Device: Placebo PBMT/sMF — The placebo PBMT/sMF will be irradiated in the lower thorax and neck areas, with the patients in supine position. PBMT/sMF application time will be 60 seconds per site. The dose used for applications during the treatment will be 0 Joules (J) per site. The sounds and signals emitted from the device as well as the information displayed on the screen will be identical, regardless of the type of treatment (active or placebo). PBMT/sMF will be applied using the direct contact method with light pressure on the skin.
  Arms: Placebo PBMT/sMF

SUMMARY:
Coronavirus disease 2019 (COVID-19) is a disease caused by a novel coronavirus called SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2). The most characteristic symptom of patients with COVID-19 is respiratory distress, leading to inability to sustain spontaneous breathing. In addition, patients with COVID-19 have dyspnea and respiratory muscle fatigue. Therefore, it is necessary to use strategies that minimize the impact of COVID-19 on the respiratory muscles, accelerating the ventilatory weaning process and optimizing the functional capacity of the involved muscles.

Over the past years, evidence has shown the effectivity of photobiomodulation therapy (PBMT) combined with static magnetic field (sMF) (PBMT/sMF) in delaying muscle fatigue, decrease in markers of inflammatory damage and oxidative stress of skeletal muscle. These effects result in an improvement in the functional capacity of the irradiated muscles by PBMT/sMF. However, do date, there is a lack of evidence regarding the effects of PBMT/sMF on the respiratory muscles.

Therefore, the irradiation of PBMT/sMF may result in improvement in the functional capacity of respiratory muscles in patients with COVID-19, accelerating the ventilatory weaning process of the patients intubated due to respiratory failure. In addition, the irradiation of PBMT/sMF may induce the increase of anti-inflammatory mediators' activity in patients with COVID-19.

Thus, the aim of this project is to investigate the effects of PBMT/sMF on respiratory muscles of patients admitted to the Intensive Care Unit (ICU) with COVID-19 using invasive mechanical ventilation.

DETAILED DESCRIPTION:
To achieve the proposed objectives it will be performed a randomized, triple-blind, placebo-controlled trial, with patients admitted to the adult ICU with COVID-19 using invasive mechanical ventilation due to respiratory failure. The patients will be randomly allocated to two treatment groups: 1. Active PBMT/sMF (MR5™ ACTIV PRO LaserShower) or Placebo PBMT/sMF (MR5™ ACTIV PRO LaserShower). The patients will be treated by a blinded therapist, and the patients will be blinded to the treatment received.

Since there are no studies in this field, initially it will be randomized 30 patients (15 patients per group) to determine the final sample size for this study.

The patients randomly allocated to the two groups will be subjected to treatment once a day, during the ICU stay, until discharge or death.

All data will be collected by a blinded assessor. The investigators will analyze:

1. Number of days hospitalized in the ICU until discharge or death.
2. Survival rate: rate of how many people survived and were discharged and how many died.
3. Muscular function of the diaphragm: the first assessment will be performed within 24 hours after the patient's intubation, the second 10 days after the first, and the third at the pre-discharge from the ICU.
4. Blood tests: baseline (admission to the ICU), 10 days after the admission, and endpoint (discharge or death).
5. Mechanical ventilation control parameters: baseline (admission to the ICU), 10 days after the admission, and endpoint (discharge or death).
6. Arterial Blood Gas Analysis: baseline (admission to the ICU), 10 days after the admission, and endpoint (discharge or death).

The data regarding the blood tests and arterial blood gas analysis will be collected directly from electronic medical record of each patients, since it is a daily hospital routine to perform these blood tests. The data will be collected by two assessors blinded to the treatment applied. The mechanical ventilation control parameters will be collected directly in the mechanical ventilator.

Statistical analysis: All the data will be analyzed by a blinded researcher not involved in data collection. The findings will be tested for their normality using the Kolmogorov-Smirnov test. Parametric data will be expressed as mean and standard deviation and non-parametric data as median and respective upper and lower limits, data can be also expressed as frequency (%). Parametric data will be analysed by two-way repeated measures analysis of variance (time vs experimental group) with post hoc Bonferroni correction. Non-parametric data will be analysed using the Friedman test and, secondarily, the Wilcoxon signed-rank test. The association between categorical variables will be analyzed using the Chi-square test or Fisher's exact test. The significance level will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the adult Intensive Care Unit with Covid-19 infection;
* Need for orotracheal intubation;
* Invasive mechanical ventilation due to respiratory failure.

Exclusion Criteria:

* Suspected patients who had a negative result of the diagnostic examination for COVID-19 infection;
* Patients positioned in pronation for more than 24 hours;
* Cancer patients;
* Pregnancy.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-09-17 (Actual); Study Completion 2020-09-17 (Actual)

PRIMARY OUTCOMES:
Time until discharge | From date of randomization until the date of discharge or date of death from any cause, whichever came first, assessed up to 20 days.
  Number of days hospitalized in the ICU until discharge or death.

SECONDARY OUTCOMES:
Survival rate | From date of randomization until the date of discharge or date of death from any cause, whichever came first, assessed up to 20 days.
  Rate of how many people survived and were discharged and how many died.
Diaphragm muscle function | 10 days after randomization and in the last test before discharge or death from any cause, whichever came first, assessed up to 20 days.
  Diaphragm thickness will be measured by ultrasound.
Platelet count | 10 days after randomization and in the last test before discharge or death from any cause, whichever came first, assessed up to 20 days.
  Platelet count will be measured by blood test.
Leukogram | 10 days after randomization and in the last test before discharge or death from any cause, whichever came first, assessed up to 20 days.
  Leukogram will be measured by blood test.
Erythrogram | 10 days after randomization and in the last test before discharge or death from any cause, whichever came first, assessed up to 20 days.
  Erythrogram will be measured by blood test.
C-reactive protein | 10 days after randomization and in the last test before discharge or death from any cause, whichever came first, assessed up to 20 days.
  C-reactive protein will be measured by blood test.
D-dimer | 10 days after randomization and in the last test before discharge or death from any cause, whichever came first, assessed up to 20 days.
  D-dimer will be measured by blood test.
Immunoglobulin G | 10 days after randomization and in the last test before discharge or death from any cause, whichever came first, assessed up to 20 days.
  Immunoglobulin G will be measured by blood test.
Immunoglobulin M | 10 days after randomization and in the last test before discharge or death from any cause, whichever came first, assessed up to 20 days.
  Immunoglobulin M will be measured by blood test.
Levels of positive end-expiratory pressure (PEEP) | 10 days after randomization and in the last test before discharge or death from any cause, whichever came first, assessed up to 20 days.
  The levels of PEEP will be measured using a mechanical ventilator.
Fraction of inspired oxygen (FiO2) | 10 days after randomization and in the last test before discharge or death from any cause, whichever came first, assessed up to 20 days.
  The levels of FiO2 will be measured using a mechanical ventilator.
Arterial partial pressure of oxygen (PO2) | 10 days after randomization and in the last test before discharge or death from any cause, whichever came first, assessed up to 20 days.
  PO2 will be measured by arterial blood gas analysis.
Arterial partial pressure of oxygen (PO2)/Fraction of inspired oxygen (FiO2) ratio | 10 days after randomization and in the last test before discharge or death from any cause, whichever came first, assessed up to 20 days.
  PO2/FiO2 ratio will be measured by arterial blood gas analysis.
Levels of tumor necrosis factor-α (TNF-α) | 10 days after randomization and in the last test before discharge or death from any cause, whichever came first, assessed up to 20 days.
  Levels of TNF-α will be measured by blood test.
Levels of vitamin D | 10 days after randomization and in the last test before discharge or death from any cause, whichever came first, assessed up to 20 days.
  Levels of vitamin D will be measured by blood test.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Tacchini, Bento Gonçalves, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] De Marchi T, Francio F, Ferlito JV, Weigert R, de Oliveira C, Merlo AP, Pandini DL, Pasqual-Junior BA, Giovanella D, Tomazoni SS, Leal-Junior EC. Effects of Photobiomodulation Therapy Combined with Static Magnetic Field in Severe COVID-19 Patients Requiring Intubation: A Pragmatic Randomized Placebo-Controlled Trial. J Inflamm Res. 2021 Jul 24;14:3569-3585. doi: 10.2147/JIR.S318758. eCollection 2021. PMID 34335043